CLINICAL TRIAL: NCT02866123
Title: Prospective Study to Evaluate Ultrasound Verification of the Correct Position of Gastric Tubes in Intensive Care
Brief Title: Verification of Correct Positioning of a Gastric Tube by Ultrasonography
Acronym: SNG echo
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Couteau-Girard 2014
Record Dates: First submitted 2016-08-04; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-07

CONDITIONS: Insertion of a Nasogastric Tube; Intubated Patient; Patients Hospitalized in the Surgery Intensive Care Unit
MeSH Terms: interventions — High-Energy Shock Waves

ARMS (1):
- patient with insertion of an NGT (Experimental)
  Interventions: Other: ultrasonography; Radiation: pulmonary radiography

INTERVENTIONS:
Other: ultrasonography
Radiation: pulmonary radiography

SUMMARY:
There are several ways to verify the correct positioning of a gastric tube. Radiography is considered the reference method. The use of ultrasonography could diminish the number of radiographies necessary. The hypothesis of this research is that gastric ultrasonography performed during insertion of the tube is a reliable examination to check the correct positioning of gastric tubes in intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Patients, or their persons of trust, in cases of coma or sedated patients) who have given informed oral consent
* All patients hospitalized in the surgery intensive care unit of Dijon CHU, who are intubated and require a gastric tube

Exclusion Criteria:

* Adults under guardianship, patients under 18 years of age
* Patients without national health insurance cover
* Pregnant women
* Wound or dressing preventing gastric ultrasonography (laparotomy is not an exclusion criterion if the dressing does not prevent ultrasonography being performed)
* result of the radiographic verification seen before the gastric ultrasonography is done

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of ultrasonography examinations validating the correct insertion of a nasogastric tube (NGT) | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France